CLINICAL TRIAL: NCT00628628
Title: Phase 2 Study of Rasburicase Administered by Two Different Schedules (Fixed Dosing vs. As Needed Dosing) in Patients at High Risk or Potential Risk for Tumor Lysis Syndrome
Brief Title: Rasburicase in Patients at Risk for Tumor Lysis Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0918
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-05

CONDITIONS: Tumor Lysis Syndrome
Keywords: Tumor Lysis Syndrome; TLS; hyperuricemia; Leukemia; Lymphoma; Acute myeloid leukemia; Chronic myelocytic leukemia; CML; lactate dehydrogenase; LDH; Myelodysplastic Syndrome; Rasburicase; Elitek™
MeSH Terms: conditions — Tumor Lysis Syndrome; Hyperuricemia; Leukemia; Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes | interventions — rasburicase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): As Needed Rasburicase .15 mg/kg IV Over 30 Minutes On Day 1. Day 2-5, once daily as needed.
  Interventions: Drug: As Needed Rasburicase
- Group B (Experimental): Fixed Dose Rasburicase .15 mg/kg IV Over 30 Minutes Daily
  Interventions: Drug: Fixed Dose Rasburicase

INTERVENTIONS:
Drug: As Needed Rasburicase — .15 mg/kg IV Over 30 Minutes On Day 1. Day 2-5, once daily as needed.
  Other Names: Elitek™
  Arms: Group A
Drug: Fixed Dose Rasburicase — .15 mg/kg IV Over 30 Minutes Daily
  Other Names: Elitek™
  Arms: Group B

SUMMARY:
Primary Objectives:

To determine the efficacy of rasburicase administered as a single dose followed by as needed dosing (investigational arm) as compared to fixed dosing for 5 days (standard treatment arm) in the treatment of patients at high risk or potential risk for tumor lysis syndrome.

Secondary Objectives:

1. To evaluate the plasma uric acid area under the curve (AUC) from baseline through 7 days
2. To evaluate the incidence of renal insufficiency and electrolyte abnormalities.
3. To determine the safety and immunogenicity of rasburicase.
4. To evaluate the cost-effectiveness of the experimental treatment (investigational arm).

DETAILED DESCRIPTION:
The Study Drug and TLS Rasburicase is designed to help decrease or prevent the high level of uric acid that may occur during the start of chemotherapy. A high level of uric acid in the blood may lead to decreased kidney function or kidney failure.

TLS occurs when high uric acid levels are caused by breakdown of tumor cells during the start of chemotherapy. The dead tumor cells can release uric acid and cause other symptoms of kidney failure, such as releasing large amounts of potassium and phosphorus (chemicals) into the blood.

Screening Tests Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study.

Your complete medical history will be recorded. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight.

Blood will be drawn (about 2 tablespoons) for routine tests. Women who are able to have children must have a negative blood (using a sample from the routine blood draw) or urine pregnancy test.

Study Groups If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. There is an equal chance of being in either group.

Group A Participants in Group A will receive rasburicase by vein, over 30 minutes, on Day 1 of Cycle 1 of chemotherapy. On Days 1-7 of Cycle 1 of chemotherapy, blood (about 2 tablespoons) will be drawn for routine tests, including a check of the level of uric acid in your blood. During Days 2-5 of Cycle 1 of chemotherapy, you will only receive rasburicase (once a day) if the levels of uric acid are high that day.

Group B Participants in Group B will receive rasburicase by vein, over 30 minutes, once a day from Days 1-5 of Cycle 1 of chemotherapy. On Days 1-7 of Cycle 1 of chemotherapy, blood (about 2 tablespoons) will be drawn for routine tests, including a check of the level of uric acid in your blood.

Both Groups Treatment with rasburicase will only be given in Cycle 1 of chemotherapy. The chemotherapy will be given at least 4 hours (up to 24 hours) after the first dose of rasburicase.

Length of Study When your blood test results show that you do not have antibodies to rasburicase, your participation in this study will be over. You will be taken off this study if the TLS gets worse or intolerable side effects occur.

This is an investigational study. Rasburicase is commercially available, but it is not FDA approved for treating TLS. It is FDA approved for pediatric patients with leukemia, lymphoma, and solid tumor cancers who are receiving anti-cancer therapy that is expected to increase the blood levels of uric acid (the result of cancer cells dying from treatment). For treating TLS in adult patients, it has been authorized for use in research only. Up to 80 evaluable patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematological malignancies (leukemia/lymphoma) at high risk or potential risk for tumor lysis syndrome. High risk: hyperuricemia of malignancy (Uric acid levels >7.5); diagnosis of very aggressive lymphoma/leukemia based on Revised European-American Lymphoma (REAL) classification; acute myeloid leukemia, chronic myelocytic leukemia (CML) in blast crisis; high grade myelodysplastic syndrome only if they have >10% bone marrow blast involvement and given aggressive treatment similar to acute myeloid leukemia (AML) (continued on #2)
2. (continued from # 1) Potential risk: diagnosis of aggressive lymphoma/leukemia based on (REAL) classification. Plus one or more of the following criteria: lactate dehydrogenase (LDH) >/= 2 x upper limit of normal (ULN); Stage III-IV disease; Stage I-II disease with at least 1 lymph node/tumor >5cm in diameter.
3. ECOG performance status 0-3
4. Life expectancy >3 months
5. Negative pregnancy test (females of child bearing potential) within </=2 weeks of rasburicase dose and use of efficient contraceptive method (both males and females). Pregnancy test may be performed on serum (HCG) or urine (HCG)
6. Signed written informed consent (approved by the Institutional Review Board/Ethics Committee) obtained prior to study entry

Exclusion Criteria:

1. Patient receiving any investigational drug for hyperuricemia within 30 days of planned first treatment with rasburicase
2. Pregnancy or lactation
3. Known history of significant allergy problem or documented history of asthma or asthmatic bronchitis
4. Known history of glucose-6-phosphate dehydrogenase deficiency
5. Known history of hemolysis and methemoglobinemia
6. Previous therapy with urate oxidase
7. Other conditions unsuitable for participation in the trial in the Investigator's opinion
8. Unwillingness to comply with the requirements of the protocol
9. Use of allopurinol within 72 hours of the study entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Vadhan-Raj S, Fayad LE, Fanale MA, Pro B, Rodriguez A, Hagemeister FB, Bueso-Ramos CE, Zhou X, McLaughlin PW, Fowler N, Shah J, Orlowski RZ, Samaniego F, Wang M, Cortes JE, Younes A, Kwak LW, Sarlis NJ, Romaguera JE. A randomized trial of a single-dose rasburicase versus five-daily doses in patients at risk for tumor lysis syndrome. Ann Oncol. 2012 Jun;23(6):1640-5. doi: 10.1093/annonc/mdr490. Epub 2011 Oct 19. PMID 22015451
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 28, 2008 to March 8, 2010. All participants were recruited in a medical clinic setting at The UT MD Anderson Cancer Center.
Pre-assignment Details: Eighty-two patients were enrolled between February 2008 and February 2010. Two patients withdrew consent and 80 patients were randomized; 40 to the Arm A and 40 to the Arm B.
Groups:
- Group A: Single Dose: As Needed Rasburicase .15 mg/kg IV Over 30 Minutes On Day 1. Day 2-5, once daily as needed.
- Group B: Daily Dose: Fixed Dose Rasburicase .15 mg/kg IV Over 30 Minutes Daily
Period: Overall Study
Arm/Group | Group A: Single Dose | Group B: Daily Dose
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Single Dose | Group B: Daily Dose | Total
Number analyzed (Participants) | 40 | 40 | 80
Age Continuous [Median (Full Range); unit: years] | 62 [27 to 82] | 58 [27 to 81] | 60 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma Uric Acid (UA) Response
Description: Plasma UA response is defined as normalization of plasma UA levels within 48 hours after the start of study drug (rasburicase) and maintaining within the normal range after the final drug infusion on day 5. Plasma samples for UA were collected at baseline before rasburicase, 4- and 24-hours post-rasburicase, and daily during treatment.
Time Frame: First cycle of chemotherapy, up to 5 days
Measure: Number; unit: participants
Arm/Group | Group A: Single Dose | Group B: Daily Dose
Number analyzed (Participants) | 40 | 40
participants | 39 | 34

ADVERSE EVENTS:
Time Frame: 2 years, 1 month
Arm/Group | Group A: Single Dose | Group B: Daily Dose
Serious Adverse Events (participants affected / at risk) | 0/40 | 2/40
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Single Dose (N=40) | Group B: Daily Dose (N=40)
Leukemia (Blood and lymphatic system disorders) | 0 | 1
Lymphoma (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Single Dose (N=40) | Group B: Daily Dose (N=40)
Methemoglobinemia (Blood and lymphatic system disorders) | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Clinical tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 3
Laboratory tumor lysis syndrome (Metabolism and nutrition disorders) | 14 | 11
Hyperuricemia (Blood and lymphatic system disorders) | 13 | 11
Hyperphosphatemia (Blood and lymphatic system disorders) | 16 | 12
Hypocalcemia (Blood and lymphatic system disorders) | 28 | 20
Hyperkalemia (Blood and lymphatic system disorders) | 1 | 1
Increased serum creatinine (Renal and urinary disorders) | 0 | 4
Renal events requiring dialysis (Renal and urinary disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No